CLINICAL TRIAL: NCT01155713
Title: A Randomized, Open-label, Multi-center, Phase I, Crossover Study to Assess the Relative Bioavailability of 2 Oral Formulations of TKI258 (CSF Capsule vs. FMI Tablet), and the Effect of Food on the Bioavailability of TKI258, in Patients With Advanced Solid Tumors
Brief Title: Bioavailability and Food Effect Study of TKI258 (CSF Capsule vs. FMI Tablet) in Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258A2116
Record Dates: First submitted 2010-06-30; First posted 2010-07-02 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2016-05

CONDITIONS: Neoplasm; Cancer; Tumors
Keywords: Neoplasms; Cancer; Tumors; Administration, oral; Capsules; CHIR258, CHIR-258, CHIR 258, TKI258, TKI-258, TKI 258,; Bioavailability,; Food
MeSH Terms: conditions — Neoplasms | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 - TKI258 - bioavailability (Experimental)
  Interventions: Drug: TKI258
- TKI258 - food effect (Experimental)
  Interventions: Drug: TKI258

INTERVENTIONS:
Drug: TKI258
  Other Names: Dovitinib

SUMMARY:
This study will evaluate the relative bioavailability of 2 oral formulations of TKI258, and the effect of food on the bioavailability of TKI258, in adult patients with advanced solid tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an advanced solid tumor which has progressed despite standard therapy, or for which no standard therapy exists
* World Health Organization (WHO) performance status ≤ 2
* Patient must meet protocol-specified laboratory values

Exclusion Criteria:

* Patients with brain cancer
* Patients who have concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study
* Patients who have not recovered from previous anti-cancer therapies
* Female patients who are pregnant, breast feeding, or not willing to use an effective method of birth control

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Determine the relative bioavailability of the final market image form of TKI258 (monohydrate tablets) as compared to the clinical service form of TKI258 (anhydrate capsules) | relative bioavailability (9 days)
Determine the effect of food on the bioavailability of TKI258 | food effect (22 days)

SECONDARY OUTCOMES:
Characterize the safety and tolerability of TKI258, including acute and chronic toxicities. | Up to 28 days after the last dose of study drug
Evaluate preliminary evidence of anti-tumor activity of TKI258 in patients with advanced solid tumors. | Every 8 weeks until progression of disease

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (4):
  - Scottsdale Healthcare/TGen Clinical Research Service TGen Clinical Research Service, Scottsdale, Arizona
  - Duke University Medical Center, Durham, North Carolina
  - Sarah Cannon Research Institute Sarah Cannon Research Instit, Nashville, Tennessee
  - University of Utah / Huntsman Cancer Institute, Salt Lake City, Utah

REFERENCES:
- See also: Results for CTKI258A2116 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=12884